CLINICAL TRIAL: NCT04124510
Title: An 12-week, Prospective, Interventional, Single-arm, Multi-centre, Phase III Study to Examine the Efficacy and Safety of Flutiform K-haler in Asthma Patients Who Are Not Adequately Controlled by Mid-doseICS/LABA DPI Treatment
Brief Title: Efficacy and Safety of Flutiform K-haler in Patients With Uncontrolled Asthma Following Mid-dose ICS/LABA DPI Therapy
Acronym: SWIFT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The Contract of K-haler products had been terminated between Mundipharma and provider. Therefore, this clinical trial was terminated early.
Sponsor: Mundipharma Korea Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FLT18-KR-301
Record Dates: First submitted 2019-09-30; First posted 2019-10-11 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brand Name: Flutiform K-haler (Experimental): Brand Name: Flutiform K-haler Generic name: Fluticasone/formoterol dosage form: oral inhalation
  Interventions: Drug: Brand Name: Flutiform K-haler

INTERVENTIONS:
Drug: Brand Name: Flutiform K-haler — Brand Name: Flutiform K-haler Generic name: Fluticasone/formoterol dosage form: oral inhalation
  Other Names: Flutiform K-haler

SUMMARY:
The purpose of this study is to evaluate the efficacy of the Asthma improvement of Flutiform K-haler after 12 weeks of treatment in patients with moderate to severe uncontrolled* asthma following mid-dose ICS/LABA DPI therapy.

DETAILED DESCRIPTION:
Asthma is a chronic inflammatory allergic disease of airway involving many cells and various media. Airway inflammation causes various symptoms of airway hypersensitivity, including repeated wheezing, dyspnea, and tightness in the chest. An estimated 300 million people worldwide suffer from asthma, and in South Korea, an estimated asthma prevalence rate for adults is approximately 5% [1]. For more effective management of asthma, Global Initiative for Asthma (GINA) guideline[2] and Korean Asthma Management Guideline for Adults [1] suggests that for patients who cannot have asthma symptoms under control with ICS (Inhaled Corticosteroid) alone, concomitant treatment of ICS/LABA is more effective than dose increase of ICS, and therefore recommends ICS combined with Long-acting β2-agonist (LABA) products. Common ICS/LABA products that are available in the Korea market including dry power inhaler (DPI) and pressured metered dose inhaler (pMDI).

It is known that small airway significantly contributes to total airway resistance, so the inflammation of the small airways could lead to the poor asthma control observed since small airways are not directly reached by inhaler's particles [3,4]. Fluticasone/formoterol (Flutiform®) shows a high fine particle fraction (FPF) of about 40% for both the ICS and the LABA components regardless the inhalation flow rate[5]. FPF of Fluticasone/formoterol is significantly higher than other ICS/LABA combinations. It is expected that small particles of fluticason/formoterol could reach to the large/small airways easier than other ICS/LABA combinations even if these ICS/LABAs shows a similar efficacy for asthma treatment. However Asthma patients can struggle to use their pMDI inhalers correctly due to the need to properly co-ordinate the press and inhale, which can worsen their asthma and lead to exacerbations.

Flutiform K-haler is the first breath-actuated inhaled corticosteroid (ICS) long-acting β2-agonist (LABA) combination aerosol inhaler for adults and adolescents. The flutiform k-haler has been designed with patients in mind, requiring only a gentle inhalation to trigger the dose release, with the aim to help patients reduce critical errors and improve long-term outcomes.

Therefore, It is expected that Flutiform K-haler prevents exacerbation and improves symptom of Asthma. Especially it will be beneficial to patients who did not response to existing ICS/LABA DPI in Korea. This study is planned to examine the efficacy and safety of Flutiform K-haler in patients who are not adequately controlled by previous mid-dose ICS/LABA DPI treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Korean asthma patients age ≥ 19 years old
2. Patients who have moderate to severe persistent asthma, as defined by GINA 2018 guideline, with ICS/LABA DPI use history
3. Patients who have uncontrolled asthma in FEV1 up to 60% and Asthma control test score < 20
4. Female subjects of child bearing potential must have a negative urine pregnancy test prior to first dose of study medication and that they must be agree to use adequate contraception during the study period
5. Patients who are able to use the inhaler
6. Patients who is willing to voluntarily sign the study consent form

Exclusion Criteria:

1. Patients who have diagnosed as clinically significant pulmonary diseases
2. Patients who have experienced life-threatening asthma within 12 months prior to screening or respiratory infection within 4 weeks prior to screening, or patients who have experienced any emergency visit or hospitalization due to acute asthma symptoms within 4 weeks prior to screening
3. Current and past smoker: Smoker defined as below

   * Current smoker: smoking history within 90 days prior to screening
   * Past smoker: smoking amount >10 pack year
4. Patients who currently are pregnant or lactating
5. Patients who are participating or going to participate in any interventional clinical trials
6. QT interval prolongation in ECG result at screening (420msec > male, 440msec > female)
7. Patients with hypersensitive to investigational products or to any component of the drug
8. Patients requiring treatment with any of the prohibited concomitant medications Use of the following medications is prohibited during the study due to drug-to-drug interaction with the study drug
9. Patients who took SPIRIVA within 3 month prior to enrollment
10. Patients who did not show previous DPI drug compliance between 70% ~130%

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2020-09-14 (Actual); Study Completion 2020-09-14 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study is the change in Asthma control test from baseline to Week 12 on treatment | Week 0, Week 12
  change in Asthma control test from baseline to Week 12 on treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kwang Ha Yoo, Principal Investigator — Konkuk University Medical Center
Locations (1):
- Konkuk University Medical Center, Seoul, South Korea